CLINICAL TRIAL: NCT00709969
Title: Open Label, Multicenter Study for Evaluation of Safety and Efficacy of Artemether-Lumefantrine Tablets (6-Dose Regimen) in African Infants and Children in the Treatment of Acute Uncomplicated Falciparum Malaria
Brief Title: Evaluation of Safety and Efficacy of Artemether-Lumefantrine Tablets in African Infants and Children With Uncomplicated P. Falciparum Malaria
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: World Health Organization (Other); Avenue Appia 20 (Unknown); CH - 1211 Geneva 27 (Unknown); Switzerland (Unknown)
Responsible Party: External Affairs, Novartis
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCOA566A2403
Record Dates: First submitted 2008-07-02; First posted 2008-07-03 (Estimated); Last update posted 2008-07-03 (Estimated); Status verified 2008-07

CONDITIONS: Plasmodium Falciparum Malaria
Keywords: Malaria; co-artemether; auditory; Plasmodium falciparum; marsh fever; remittent fever; artemether; artemisinins; lumefantrine; child; infant; Africa
MeSH Terms: conditions — Malaria, Falciparum; Malaria | interventions — Artemether, Lumefantrine Drug Combination

ARMS (1):
- 1 (Experimental): Artemether-lumefantrine
  Interventions: Drug: Artemether-lumefantrine

INTERVENTIONS:
Drug: Artemether-lumefantrine — 20mg artemether and 120 mg lumefantrine, tablet, dose based on body weight, 3 days treatment 5 - < 10kg (BWG 1) = 6 doses of 1 tablet / 10 - < 15kg (BWG 2) = 6 doses of 1 tablet / 15 - ≤ 25kg (BWG 3) = 6 doses of 2 tablets
  Other Names: Coartem®, Riamet®, co-artemether

SUMMARY:
This study will assess the safety and efficacy of artemether-lumefantrine tablets (6-dose regimen) in African infants / children with acute uncomplicated falciparum malaria.

ELIGIBILITY:
Inclusion Criteria:

* male or female weighing ≥ 5kg and ≤ 25kg
* P. falciparum parasitemia between 1,000 and 100,000 parasites/mm3
* with confirmed diagnosis of uncomplicated malaria caused P. falciparum parasite

Exclusion Criteria:

* complicated malaria
* ingestion of various antimalarial drugs, or other drugs influencing cardiac function in the previous 4 weeks before study entry to 8 weeks
* severe anaemia
* severe malnutrition
* malaria due to other than P. falciparum

Other protocol-defined inclusion/exclusion criteria may apply

Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2002-07; Study Completion 2003-02 (Actual)

PRIMARY OUTCOMES:
Adverse events, SAEs; hematology and biochemistry parameters; electrocardiogram; urine values; vital signs; physical neurological examinations; and neurological examinations | 28 days

SECONDARY OUTCOMES:
Proportion of patients free of parasites at 7, 14 and at 28 days
Time to clearance from parasites (asexual forms)
Time to clearance of fever
Time to clearance of gametocytes (parasite sexual forms)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — Novartis Pharmaceuticals
Locations (3):
- Kemri-Wellcome Trust Programme, Kilifi, Kenya
- University College Hospital Malaria Research Laboratories Institute for Advance Medical Research and Training, Ibadan, Nigeria
- Muhimbili University College of Health Sciences Department of Parasitology and Medical Entomology, Box 65011, Dar es Salaam, Tanzania

REFERENCES:
- [Derived] Falade CO, Ogunkunle OO, Dada-Adegbola HO, Falade AG, de Palacios PI, Hunt P, Virtanen M, Oduola AM, Salako LA. Evaluation of the efficacy and safety of artemether-lumefantrine in the treatment of acute uncomplicated Plasmodium falciparum malaria in Nigerian infants and children. Malar J. 2008 Nov 27;7:246. doi: 10.1186/1475-2875-7-246. PMID 19038036